CLINICAL TRIAL: NCT02755363
Title: Evaluation of the Immediate Effects of Osteopathic Techniques on Plethysmographic Measurement of Residual Volume in Patients With Severe Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Osteopathic Techniques on Residual Volume in Severe Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: WarsawMU
Record Dates: First submitted 2016-04-19; First posted 2016-04-28 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: COPD
Keywords: COPD; residual volume; osteopathy; hyperinflation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- osteopathic manual therapy (OMT group) (Active Comparator): patients who will undergo manual osteopathic therapy.
  Interventions: Other: osteopathic manual therapy
- control group (C group) (Placebo Comparator): patients who will undergo manual therapy not aimed to decrease hyperinflation.
  Interventions: Other: control group

INTERVENTIONS:
Other: osteopathic manual therapy — * suboccipital decompression - atlanto-occipital joint relaxation technique.
  * deep cervical fascia release - the technique aims to improve mobility of the first and second ribs during expiration and to relaxation of the vagus and phrenic nerve course area.
  * thoracic lymphatic pump with activation is designed to reduce the tension of mediastinal structures, improve lymphatic flow, and thus reduce the breathing resistance.
  * stretching the diaphragm in order to relax and reduce adhesion within the fascial system between the diaphragm and abdominal organs.
  Arms: osteopathic manual therapy (OMT group)
Other: control group — * manual mobilization techniques of the slides in the shoulder joint toward the front, rear and bottom.
  * manual techniques to increase range of motion in the shoulder joints using the patient's breathing manoeuvres.
  Arms: control group (C group)

SUMMARY:
The purpose of this study is to determine whether the selected osteopathic techniques have a positive impact on the residual volume decrease in patients with chronic obstructive pulmonary disease with severe and very severe airflow limitation in comparison to the manual therapy not aimed to decrease hyperinflation (placebo).

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterized by progressive and not fully reversible airflow limitation in the bronchi.

Hyperinflation is one of the most important pathophysiological mechanisms responsible for shortness of breath in COPD patients. Hyperinflation may be assessed in body pletysmography in which residual volume (RV) and total lung capacity (TLC) are measured. These parameters are considered to precisely reflect the degree of hyperinflation. In patients with COPD, an increased breathing frequency, e.g. during exercise or disease exacerbation, leads to dynamic hyperinflation which further increases shortness of breath.

The treatment of COPD includes smoking cessation, drug therapy, home oxygen therapy and rehabilitation. The disease is chronic, progressive and ultimately leads to premature death, so every new therapeutic option is a point of interest. In the recent years, there have been a few reports on the positive effects of osteopathic techniques on pulmonary function tests in patients with COPD. Osteopathy is a new area of healthcare, in which manual techniques are used to assess neuro-musculoskeletal performance and to optimize its function.

STUDY OBJECTIVE the assessment of the influence of selected osteopathic techniques on RV in patients with COPD (III, IV degree of airway obstruction according to Global Initiative for Chronic Obstructive Lung Disease - GOLD).

MATERIAL

The patients will be recruited from an outpatient clinic and randomly assigned to 2 groups:

* group of osteopathic manual therapy (OMT group) - 10 patients - who will undergo 25 minutes of manual osteopathic therapy;
* control group (C group)- 10 patients - who will undergo 25 minutes of manual therapy not aimed to decrease hyperinflation, as placebo.

Then, after a period of two-three weeks patients will be crossed over between the groups.

METHODS Spirometry to assess forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) and body pletysmography with the measurement of RV will be performed before and 10 minutes after the manual therapy session.

Manual therapy directed at the normalization of the autonomic nervous system (inhibition of the sympathetic nervous system) and at the improvement of chest wall mobility will be applied. The techniques are painless for the patient. In both investigated groups, all the techniques will be applied in supine position, after daily inhaled medication intake.

The techniques to be applied in the OMT group include:

* suboccipital decompression - it is based on the pressure of suboccipital muscles with fingers of the therapist at the base of the skull.
* deep cervical fascia release - the therapist will move the thumb on the neck of the patient from cranium in the caudal direction over sternocleidomastoid, scalene, trapezius muscles.
* thoracic lymphatic pump with activation is - the therapist manually supports the breathing rhythm of the patient by the compression and decompression of the sternum effecting in the sterno-costal joints relaxation and intensification of the lymph flow of in the lymphatic thoracic duct. The impact on the thoracic duct is carried out by the rhythmic pressure differences while breathing and supported with hands of the therapist.
* stretching the diaphragm - the technique relies on manual catch by 10, 11 and rib cartilage, which will be held in the inspiratory direction during exhalation of the patient.

The therapist will decide when the subsequent techniques will be terminated basing on the improvement of the flexibility and mobility of the treated area evaluated by palpation.

The techniques to be applied in the C group include:

* manual mobilization techniques of the slides in the shoulder joint toward the front, rear and bottom.
* manual techniques to increase range of motion in the shoulder joints using the patient's breathing manoeuvres.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of COPD in accordance with GOLD,
* post-bronchodilator FEV1 < 50% of predicted value,
* smoking history of ≥ 10 pack-years,
* the ability to remain in supine position for at least 25 minutes.

Exclusion Criteria:

* exacerbation in the past 6 weeks,

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Lung function tests (mainly residual volume) before and after selected osteopathic techniques in patients with COPD (III, IV degree of airway obstruction according to GOLD). | 40 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Górska, PhD, MD, Principal Investigator — WMU
Locations (1):
- Departament of Internal Medicine, Pneumonology and Allergology, Warsaw Medical University, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes